CLINICAL TRIAL: NCT05757284
Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Development of a Diagnostic Set for Patients With LLL
Brief Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Aim 3
Acronym: EvaLymph-Leg3
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Nij Smellinghe Hospital Drachten (Unknown)
Responsible Party: Principal Investigator, Tessa De Vrieze, Dr., KU Leuven
Other Study IDs: s66033-aim3
Record Dates: First submitted 2023-02-07; First posted 2023-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lower Limb Lymphedema
Keywords: severity score; diagnostic set

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with unilateral or bilateral, primary or secundary LLL
  Interventions: Diagnostic Test: Lower Limb Lymhedema assessment
- healthy controls
  Interventions: Diagnostic Test: Lower Limb Lymhedema assessment

INTERVENTIONS:
Diagnostic Test: Lower Limb Lymhedema assessment — assessessment with the selected measurement methods showing sufficient reliability and feasibility in the patient group with LLL from aim 1:NCT05269264. Measurement will occur at the genital/midline region, and on both legs/ feet.

SUMMARY:
The current best practice is a three-stage classification consensus guideline as published by the International Society of Lymphology (ISL). Severity of lymphedema is however not only determined by presence of pitting (which is the phenomenon when the swollen area has a dimple (or pit) after you press it for 5 to 10 seconds) and presence of adipose tissue or not, but is also determined by the volume of the edema, a quantification of the condition of the skin and the location/expansion of the edema over the body. Currently a severity score considering these different aspects does not exist. Although there is consensus that the ISL staging systems is a necessary part of the diagnosis of lymphedema, it gives not enough information about the severity of the lymphedema. A more detailed and comprehensive classification system applicable for primary and secondary lymphedema and considering multiple edema characteristics, remains to be formulated.

The researchers objective in this study is to develop a diagnostic set, including a 'severity score', for patients with LLL.

ELIGIBILITY:
Inclusion Criteria:

Patient group

* Unilateral or bilateral, primary or secondary LLL
* Objective diagnosis of lymphedema: ≥ 5% volume difference between both legs OR ≥ 2 minor/ 1 major criteria on lymphoscintigraphy OR presence of ICG dermal backflow
* Age ≥ 18 years
* Able to read, understand and speak Dutch

Healthy controls

- Age, gender & BMI-matched healthy controls

Exclusion Criteria:

* Pregnant participants
* Presence of chronic venous insufficiency C4, C5, C6; deep venous thrombosis; post-thrombotic syndrome
* Presence of skin infections of wounds at the level of the lower limbs at the moment of inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with LLL will be recruited in the center for lymphedema in UH Leuven in Belgium and in the center for lymphedema in Nij Smellinghe Hospital in Drachten in the Netherlands.
  Healthy volunteers, both in Belgium as well as in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of measurement methods (resulted from aim 1:NCT05269264) in diagnosing unilateral and bilateral LLL | During the recruitment period (up to 1 year), patients are scheduled for only 1 visit with duration of +/- 1 hour (cross-sectional design)
  all patients with LLL and all healthy controls will be assessed with the selected measurement methods showing sufficient reliability and feasibility in the patient group with LLL from aim 1. Measurement will occur at the genital/midline region, and on both legs/ feet.
Specificity of measurement methods (resulted from aim 1:NCT05269264) in diagnosing unilateral and bilateral LLL | During the recruitment period (up to 1 year), patients are scheduled for only 1 visit with duration of +/- 1 hour (cross-sectional design)
  all patients with LLL and all healthy controls will be assessed with the selected measurement methods showing sufficient reliability and feasibility in the patient group with LLL from aim 1. Measurement will occur at the genital/midline region, and on both legs/ feet.
Diagnostic accuracy of measurement methods (resulted from aim 1:NCT05269264) in diagnosing unilateral and bilateral LLL | During the recruitment period (up to 1 year), patients are scheduled for only 1 visit with duration of +/- 1 hour (cross-sectional design)
  all patients with LLL and all healthy controls will be assessed with the selected measurement: methods showing sufficient reliability and feasibility in the patient group with LLL from aim 1. Measurement will occur at the genital/midline region, and on both legs/ feet.
  To determine diagnostic accuracy of the diagnostic methods, in a first phase, data will be analysed using Receiver Operating Characteristic (ROC) curves and by calculation the area under the curve (AUC) for each individual evaluation method resulting from aim 1.
  Sensitivity and specificity values will be compared, and for each measurement method, the AUC (or C-statistic) will be considered. Also prognostic values and likelihood ratios will be calculated of the individual measurement methods.
  Lastly, to investigate discriminant validity, measurement outcomes of the patients with LLL will be correlated to the measurement outcomes of the healthy controls.
Development of a severity grading score for unilateral and bilateral LLL | During the recruitment period (up to 1 year), patients are scheduled for only 1 visit with duration of +/- 1 hour (cross-sectional design)
  a meeting with the international expert panel will be organized to achieve consensus regarding the measurement methods that should be performed to compile a severity score. Secondly, of all these separate measurement methods, percentiles (20, 40, 60, 80) will be calculated from the data of our study sample for this aim, serving as reference cut-off values. Consequently, 5 'severity' ranges will be presented that will correspond to a severity subscore between 0-5 for each measurement outcome. Lastly, a total severity score will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Tessa De Vrieze, Dr., Principal Investigator — KU Leuven
Locations (2):
- University Hospitals of Leuven, Leuven, Belgium
- Nij Smellinghe Hospital, Drachten, Netherlands